CLINICAL TRIAL: NCT05445739
Title: The Effect of an Online Exercise Course on the Increase of Elders' Regular Exercise Intention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202205111RINC
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-06

CONDITIONS: Elderly; Exercise Training
Keywords: exercise; older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The effect of an online exercise course on the increase of elders' regular exercise intention (Other): The effect of an online exercise course on the increase of elders' regular exercise intention.
  Interventions: Behavioral: The effect of an online exercise course on the increase of elders' regular exercise intention

INTERVENTIONS:
Behavioral: The effect of an online exercise course on the increase of elders' regular exercise intention — The intervention of an online exercise course which 2 days a week for 4 weeks to increase the elders' regular exercise intention.

SUMMARY:
The effect of an online exercise course on the increase of elders' regular exercise intention.

DETAILED DESCRIPTION:
This project expects that after the four-week exercise course intervention, the elderly can increase their knowledge about exercise and experience the benefits of exercise, enhance the intention of the elderly to exercise regularly, and reduce the chance of the elderly falling due to muscle loss and causing related diseases.

ELIGIBILITY:
Inclusion Criteria:

* The patients from outpatient clinic for elderly health examination.

Exclusion Criteria:

* The elderly who has severe hearing impairments.
* The elderly who has severe visual impairments.
* The elderly who has severe health problems.
* The elderly who need to be quarantined.
* The elderly who is living alone.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the survey of questionnaire | Baseline, within 2 weeks after the end of the intervention
  Change from baseline of exercise intention on the survey of questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Kun-Pei Lin, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: How to be Successful Aging — https://www.cgmh.org.tw/cgmn/cgmn_file/0710001.pdf
- See also: Epidemiology of Sarcopenia among Community-Dwelling Elderly in Taiwan — https://doi.org/10.6320/fjm.2014.18(3).04
- See also: Gender differences in the relationships among leisure-time physical activities, sedentary behaviors, and Health-Related Quality of Life for older adults in Taipei metropolitan area — https://doi.org/10.6288/tjph.202012_39(6).109100
- See also: Review: Sarcopenia and Frailty — https://doi.org/10.6314/jimt.2014.25(3).01
- See also: Study of the Promotive Strategies and Interventive Model for Physical Activity in Community — https://doi.org/10.6222/pej.4103.200809.0801
- See also: Effects of Physical Activity Programs Intervention on Physical Activity and Exercise Self-Efficacy of Community Residents — https://hdl.handle.net/11296/q3stcs
- See also: A Research in Relationship between Health Condition Awareness, Attitudes toward Exercises and Exercising Behaviors: A case study of Administrative Personnel of National Taitung University — https://hdl.handle.net/11296/q6dy55
- See also: A study on the regular behavior of exercise and the related factors in elementary school students — https://doi.org/10.6222/pej.0029.200009.1908
- See also: The concept and practice of physical activity intervention in lifestyle — https://doi.org/10.6223/qcpe.2303.200909.1902
- See also: Prevention and care of sarcopenia in the elderly — https://nursing.tzuchi.com.tw/images/pdf/14-2/b4.pdf
- See also: Introduction to sarcopenia — https://www.airitilibrary.com/Publication/alDetailedMesh?DocID=P20090727001-201504-201504300016-201504300016-103-107&PublishTypeID=P001
- See also: Using Extension of the Technology Acceptance Model to the Study about Older People's Willingness to Use the Exergame — https://www.airitilibrary.com/Publication/alDetailedMesh1?DocID=U0078-0510202013411841
- See also: Factors to regular exercise for the community elderly — https://www.airitilibrary.com/Publication/alDetailedMesh1?DocID=U0118-0807200916274292